CLINICAL TRIAL: NCT07136688
Title: A Randomized Control Trial of Transcutaneous Tibial Nerve Stimulation for Neurogenic Bladder in the Pediatric Population
Brief Title: Tibial Nerve Stimulation for Pediatric Spina Bifida Neurogenic Bladder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Argyrios Stampas, MD, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS- 24-1198
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Neurogenic Bladder Due to Spina Bifida
Keywords: spinal cord injury (SCI); transcutaneous tibial nerve stimulation (tTNS)
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Stamobil electric stimulator (Experimental)
  Interventions: Device: Stamobil electric stimulator
- sham tTNS device (Sham Comparator)
  Interventions: Device: sham tTNS device

INTERVENTIONS:
Device: Stamobil electric stimulator — The electric stimulation protocol will use stimulation frequency of 20 Hz and pulse width of 200ms in continuous mode for 30 minutes daily. The goal is daily use of tTNS for 4 weeks , 5 days per week.
  Arms: Stamobil electric stimulator
Device: sham tTNS device — The electric sham stimulation protocol will use sham stimulation (low intensity) for 30 minutes daily, for 4 weeks , 5 days per week
  Arms: sham tTNS device

SUMMARY:
The purpose of this study is to determine the safety, feasibility, and compliance of a daily home transcutaneous tibial nerve stimulation (tTNS) protocol in children with chronic neurogenic bladder (NB) provided by self or caregiver for 4 weeks and to estimate the efficacy of tTNS

ELIGIBILITY:
Inclusion Criteria:

* chronic neurogenic bladder
* Spina Bifida diagnosis
* Use of overactive bladder medication(s)
* Stable bladder medications for ≥ 3 months

Exclusion Criteria:

* Progressive SCI (ex: transverse myelitis, polio, etc.)
* Other lower urinary tract pathology or surgery
* 2+ pitting edema in the legs that does not resolve
* Known peripheral neuropathy or injury to the path of the tibial nerve
* Cancer in the tibial nerve pathway and/or lower urinary tract
* Inability to elicit the motor response with electric stimulation
* Inability to complete the tTNS proficiency checklist (guardians)
* Non-English speaking (guardians)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-04-11 (Estimated); Study Completion 2027-08-11 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by the number of adverse events | from start of trial to end of trial (4 weeks after start)
Feasibility as assessed by the satisfaction surveys | end of study (4 weeks after baseline)
  This is an 8 item questionnaire and each is scored from 1(strongly disagree) to 5(strongly agree) for a maximum score of 40, higher score indicating greater satisfaction .
Compliance of tTNS usage as assessed by the percent of sessions where toe flexion was elicited | from start of trial to end of trial (4 weeks after start)
  This will be reported in the TTNS log
Compliance of tTNS usage as assessed by the average current where toe flexion was elicited | from start of trial to end of trial (4 weeks after start)
  This will be reported in the TTNS log
Compliance of tTNS usage as assessed by percentage of sessions that bladder medications were taken | from start of trial to end of trial (4 weeks after start)
  This will be reported in the TTNS log
Satisfaction as assessed by the survey | end of study (4 weeks after baseline)
  This will measure the likelihood of tTNS preference over anticholinergic medication use
  This is an 8 item questionnaire and each is scored from 1(strongly disagree) to 5(strongly agree) for a maximum score of 40, higher score indicating greater satisfaction .

SECONDARY OUTCOMES:
Percentage of participants that are able to reduce their overactive bladder (OAB) medications | end of study (4 weeks after baseline)
percent dose reduction (mg ) achieved | end of study (4 weeks after baseline)
Change in maximum detrusor pressure (Max Pdet (cmH20)) as assessed by the Urodynamic study (UDS) | week 0, week 4
Presence of Detrusor overactivity (DO) as assessed by the Urodynamic study (UDS) | week 0
Presence of Detrusor overactivity (DO) as assessed by the Urodynamic study (UDS) | Week 4
Change in maximum volume (mL) that bladder can hold before voiding or discomfort as assessed by the Urodynamic study (UDS) | Week 0, Week 4
Presence of bladder leak as assessed by the Urodynamic study (UDS) | Week 0
Presence of bladder leak as assessed by the Urodynamic study (UDS) | Week 4
Change in bladder sensation as assessed by the Urodynamic study (UDS) | Week 0, Week 4
  volume infused (mL) at 1) time of reported first sensation of filling, 2) time of reported urgency/desire to void, & 3) time of reported discomfort
Change in detrusor compliance as assessed by the Urodynamic study (UDS) | Week 0, Week 4
  reported as change in bladder volume divided by change in bladder pressure.
Number of incontinence episodes as reported in the voiding diary | from start of trial to end of trial (4 weeks after start)
Frequency of catheterization as reported in the voiding diary | from start of trial to end of trial (4 weeks after start)
Volumes of catheterization as reported in the voiding diary | from start of trial to end of trial (4 weeks after start)
Change in bladder symptoms as assessed by the Neurogenic Bladder Symptom Score (NBSS) | Week 0, Week 4
  This is a 24 item questionnaire that is scored from 0 (no symptoms) to 4 (worst symptoms), maximum score of 96 with higher values indicating greater symptom burden
Change in bowel function as assessed by the Neurogenic Bowel Dysfunction Score (NBDS) | Week 0, Week 4
  This is a 10 item questionnaire that is scored from 0 (very minor ) to greater than or equal to 14(severe), maximum score range of 0-47 with higher scores indicating worse outcome
Change in general physical and mental health status as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire for Global Health | Week 0, Week 4
  This is a 10 item questionnaire. The measure yields two standardized summary scores: Global Physical Health (GPH) and Global Mental Health (GMH).Each summary score is calculated based on 4 items from the questionnaire and is converted to a T-score using the PROMIS scoring manual. T-scores have a mean of 50 and standard deviation of 10, based on the U.S. general population. Higher T-scores indicate better health.

CONTACTS AND LOCATIONS:
Overall Officials: Argyrios Stampas, MD, MS, Principal Investigator — The University of Texas Health Science Center and Houston
Locations (1):
- The University of Texas Health Science Center and Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No